CLINICAL TRIAL: NCT06970275
Title: A Multicentric, Observational, Post-marketing, Registry Study to Assess the Correlation of High-resolution Specimen PET-CT Imaging, Using the XEOS AURA 10 PET-CT, With the Histopathology Results and Long-term Outcome of Patients Undergoing Resective Cancer Surgery.
Brief Title: To Assess the Correlation of High-resolution Specimen PET-CT Imaging, Using the XEOS AURA 10 PET-CT, With the Histopathology Results and Long-term Outcome of Patients Undergoing Resective Cancer Surgery.
Acronym: PETRiS
Status: Recruiting | Type: Observational
Sponsor: XEOS Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: PETRiS
Record Dates: First submitted 2025-04-25; First posted 2025-05-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancers; Breast Cancer; Head and Neck Cancer; Cancer
Keywords: PET-CT; Registry; Imaging; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

SUMMARY:
This registry study aims to evaluate the effectiveness and clinical impact of specimen PET-CT imaging by analyzing the correlation between specimen PET-CT images, intraoperative interpretations, and histopathological findings. Additionally, it assesses how these imaging insights influence clinical decision-making and long-term patient outcomes. Through this comprehensive analysis in a real-world setting, the study seeks to generate valuable insights that can enhance specimen evaluation processes and ultimately improve patient care.

ELIGIBILITY:
Inclusion Criteria :

All patients that were scheduled for resective surgery and for whom successful high-resolution PET-CT imaging was performed on their resected specimens using the AURA 10 PET-CT. Successful imaging means that the image contains at least a portion of the primary tumor, the radiotracer injection was correctly executed and there were no technical issues that lead to an uninterpretable PET-CT image. Or all patients that are scheduled for resective surgery and for whom high-resolution PET-CT imaging will be performed on their resected specimens using the AURA 10 PET-CT.

Patients willing to provide informed consent for use of their relevant medical records. For retrospectively included patients with no further Long-Term Follow-Up (LTFU) data collection, a notification will be sent.

Exclusion Criteria:

* Under the age of 18 years at the time of resective surgery.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are routinely scheduled or underwent resective surgery and for whom high-resolution PET-CT imaging is or was performed on their resected specimens, using the AURA 10 PET-CT, may participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2031-01-15 (Estimated); Study Completion 2031-01-15 (Estimated)

PRIMARY OUTCOMES:
To assess the correlation between the specimen PET-CT images and final histopathological examination of the specimen. | Perioperative
  The concordance rate between the specimen PET-CT images and final histopathological examination of the specimen.

SECONDARY OUTCOMES:
To assess the correlation between the intra-operative interpretation of specimen PET-CT images and histopathological examination of the specimen and its impact on clinical decision-making. | Perioperative
  The concordance rate between the specimen PET-CT image interpretation and histopathological examination of the specimen. This will include sensitivity, specificity, positive predictive value, and negative predictive value of the intra-operative interpretation of specimen PET-CT images compared to final histopathological examination.
  The concordance rate of the clinical decisions made based on specimen PET-CT images with the clinical decisions supported by final histopathological examination (e.g. additional resection during surgery, follow-up treatment strategy, etc).
To assess the correlation between long-term follow-up clinical outcome and specimen PET-CT imaging findings. | From surgery to 3 years long term follow-up
  The incidence of biochemical, local, regional and distant recurrence rate at 1, 2 and 3 years of follow-up.
  The measurement of functional outcome at 1, 2 and 3 years of follow-up.
To evaluate the influence of neoadjuvant treatment (NAT) on PET radiotracer uptake in specimen PET-CT imaging. | Perioperative
  The measurement of PET radiotracer uptake (in MBq/mL) in specimen PET-CT images, comparing patients with different neoadjuvant treatments and those who did not receive neoadjuvant treatment.
To investigate whether preoperatively available information (such as tumor subtype, anatomical location, tumor biology, size, grade or TNM classification) as well as intra-operatively available information influence specimen PET-CT images. | Perioperative
  The measurement of PET-tracer uptake (in MBq/mL) in specimen PET-CT images, comparing patients with various preoperatively available characteristics, as well as intra-operatively available information.
To investigate whether preoperatively available information (such as tumor subtype, anatomical location, tumor biology, size, grade or TNM classification) as well as intra-operatively available information influence specimen PET-CT images. | Perioperative
  The measurement of electron density (in Hounsfield Units (HU)) in specimen PET-CT images, comparing patients with various preoperatively available characteristics, as well as intra-operatively available information.
To investigate the influence of different PET radiotracers, activity, physiological parameters and imaging parameters on PET-radiotracer uptake and image quality in specimen PET-CT images. | Perioperative
  The measurement of radiotracer uptake (in MBq/mL) in specimen PET-CT images, comparing the uptake levels and patterns across different PET radiotracers. This will assess whether the type of PET-radiotracer used leads to significant differences in the intensity or distribution of radiotracer uptake in the PET-CT specimen images.
To investigate the influence of different PET radiotracers, activity, physiological parameters and imaging parameters on PET-radiotracer uptake and image quality in specimen PET-CT images. | Perioperative
  The assessment of PET image quality (e.g. signal to noise ratio) in relation to PET radiotracer activity. This will involve evaluating how changes in radiotracer activity impact image quality and identifying the optimal activity for improving the PET-CT specimen imaging workflow.
To investigate the influence of different PET radiotracers, activity, physiological parameters and imaging parameters on PET-radiotracer uptake and image quality in specimen PET-CT images. | Perioperative
  The assessment of PET image quality (e.g. signal to noise ratio) in relation to physiological parameters (e.g. uptake time). This will involve evaluating how changes in these parameters impact image quality and identifying the optimal parameters for improving the specimen PET-CT imaging workflow.
To investigate the influence of different PET radiotracers, activity, physiological parameters and imaging parameters on PET-radiotracer uptake and image quality in specimen PET-CT images. | Perioperative
  The assessment of PET image quality (signal to noise ratio) in relation to imaging parameters (decay time). This will involve evaluating how changes in these parameters impact image quality and identifying the optimal parameters for improving the specimen PET-CT imaging workflow.
To assess the safety profile of PET-CT imaging procedures. | From surgery to 3 years long term follow-up
  The incidence of related (serious and non-serious) adverse events following the specimen PET-CT imaging procedure, including the severity, type, and frequency and relationship (possible, probable, causal relationship).

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Maria Middelares, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided